CLINICAL TRIAL: NCT06246539
Title: Impact of a Virtual Reality-based Mindfulness Program on Clinician Wellness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Steven Bird, Professor of Emergency Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00001606
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Wellness, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - VR Mindfulness (Experimental): The intervention group will be given the VR headset for their unrestricted use over the 12 week intervention period. The VR headset is exceptionally easy and intuitive to use. Each participant will have the choice of 20 "locations" in which to use the mindfulness-based program. Each of the 20 locations/programs are different. They range in length from 5 minutes (introductory) to 20 minutes.
  Interventions: Behavioral: VR mindfulness
- Control (No Intervention): The control arm will not have any intervention. However, at the conclusion of the study, all participants from the Control group will be given the VR intervention

INTERVENTIONS:
Behavioral: VR mindfulness — VR-based mindfulness
  Arms: Intervention - VR Mindfulness

SUMMARY:
Burnout shares symptoms with anxiety and depression. While there is no single intervention for burnout, there are validated interventions (which are amenable to virtual reality (VR)) for anxiety and depression. UMassMemorial data from the Professional Well-Being Academic Consortium show that MD burnout and distress has increased since 2020. The investigators believe providing clinicians with a unique tool (VR) will be a feasible and efficacious way to tackle distress. It is known that only 1% of our MDs have done mindfulness training but nearly 50% are interested in doing so. Therefore, a self-administrable, interactive mindfulness program delivered over VR has great potential to reach clinicians who want to practice a more active form of mindfulness at a time convenient to them. The results of the study will provide preliminary evidence to determine if a take-home VR mindfulness program decreases clinician stress.

DETAILED DESCRIPTION:
Cohorts 1 will be the intervention group Cohorts 2 will be the controls. Study endpoints include results from the following questionnaires:

1. PROMIS - Short Form Anxiety (8 questions)
2. PROMIS - Short Form Depression (8 questions)
3. Perceived Stress Scale (10 questions)
4. Connor-Davidson Brief Resilience Scale (10 questions)
5. System Usability Scale (10 questions)

The intervention is a 12-week mindfulness-based VR intervention.

Cohort 1 will complete the questionnaires 1-4 at baseline (just before the intervention). They will be sent twice weekly reminders to use the VR for the duration of the 12-week intervention. After 12 weeks Cohort 1 will retake questionnaires 1-4 and take questionnaire 5, while Cohort 2 will then take questionnaires 1-4 and be provided the VR headsets. After another 12 weeks, Cohort 1 will take questionnaires 1-4 and be done with the study, while Cohort 2 will take questionnaires 1-5. After 12 more weeks, Cohort 2 will take questionnaires 1-4 and be done with the study.

ELIGIBILITY:
Inclusion Criteria:

* physician or APP employed by the Medical Group

Exclusion Criteria:

* Not willing to receive 2 texts per week

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS - anxiety | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the intervention group at 12 and 24 weeks to their baseline.
  PROMIS Short Form - anxiety scale. Scores of 8-40; Higher is a worse outcome.
PROMIS - anxiety | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the control group at 12 and 24 weeks to their baseline.
  PROMIS Short Form - anxiety scale. Scores of 8-40; Higher is a worse outcome.
PROMIS - Depression | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the intervention group at 12 and 24 weeks to their baseline.
  PROMIS Short Form - Depression scale. Scores of 8-40; Higher is a worse outcome.
PROMIS - Depression | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the control group at 12 and 24 weeks to their baseline.
  PROMIS Short Form - Depression scale. Scores of 8-40; Higher is a worse outcome.
Resiliency | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the intervention group at 12 and 24 weeks to their baseline.
  Connor-Davidson Resiliency Scale. Scores of 0-40; Higher score is better.
Resiliency | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the control group at 12 and 24 weeks to their baseline.
  Connor-Davidson Resiliency Scale. Scores of 0-40; Higher score is better.
Stress scale | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the intervention group at 12 and 24 weeks to their baseline.
  Perceived Stress Score. Scores of 0-40; Higher score is worse.
Stress scale | at baseline, after 12 weeks, then after another 12 weeks. We will compare results of the control group at 12 and 24 weeks to their baseline.
  Perceived Stress Score. Scores of 0-40; Higher score is worse.
Usability | after 12 weeks we will dertermine the usability of the VR intervention in the intervention group
  Usability scale. Scores of 10-50; Higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bird, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMassMemorial Health Care, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No